CLINICAL TRIAL: NCT00918242
Title: Assessment of Occult CAD: Premature CAD Sibling Study (PreCASS)
Brief Title: Prevalence of Coronary Artery Disease in the Siblings of Premature Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Korean Society of Lipidology and Atherosclerosis (Unknown)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Yonsei University, Yonsei University
Other Study IDs: 20090616
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; computed tomography; prevalence of coronary artery disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this prospective study is to investigate the prevalence of coronary artery disease using computed tomography with family history of premature coronary heart disease

ELIGIBILITY:
Inclusion Criteria:

* within 1 year
* the siblings of premature coronary heart disease (male<55years old, female<65yeasrs old: Framingham Heart Study) patients admitted relevant hospital

Exclusion Criteria:

* Documented coronary heart disease
* experienced adverse events with relevant treatment
* contraindicated with beta-blockers
* Any woman of childbearing potential who is pregnant, seeking to become pregnant or suspects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the siblings of premature coronary heart disease (male<55years old, female<65yeasrs old: Framingham Heart Study) patients admitted relevant hospital within 1 year
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
evaluation of prevalence to coronary artery disease using CT | within 2 weeks from CT scanning

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, MD, PhD, Principal Investigator — Cardiology Division, Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Arad Y, Spadaro LA, Goodman K, Newstein D, Guerci AD. Prediction of coronary events with electron beam computed tomography. J Am Coll Cardiol. 2000 Oct;36(4):1253-60. doi: 10.1016/s0735-1097(00)00872-x. PMID 11028480